CLINICAL TRIAL: NCT05311306
Title: A Non-interventional, Multi-centre Study to Investigate the Change in Clinical and Patient-reported Outcomes in Moderate to Severe COPD Patients Treated With TRIXEO (Budesonide / Glycopyrronium / Formoterol) Under Real-life Conditions
Brief Title: REported Outcomes in COPD With Trixeo in Real worlD in Germany
Acronym: RECORD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00037
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by persistent respiratory symptoms (including breathlessness, cough, and sputum production), which has a substantial impact on health-related quality of life (HRQoL). Medical treatment of COPD aims to reduce these symptoms, reduce exacerbations, and improve patients' ability to perform exercise and daily activities. TRIXEO is a triple therapy indicated as a maintenance treatment in adult patients with moderate-to-severe COPD who are not adequately treated by a combination of an inhaled corticosteroid and a long-acting beta2-agonist or combination of a long-acting beta2-agonist and a long-acting muscarinic antagonist.

The RECORD study is a prospective, non-interventional study to be conducted in the United Kingdom (UK) and Germany. The study aims to generate data to describe the real world effectiveness of TRIXEO for patients with COPD who receive TRIXEO in routine clinical practice. It also aims describe patients HRQoL, physical activity and treatment satisfaction, and will explore patients' sleep quality and adherence to inhalers in the real-world. This data may provide important information for practicing physicians.

The study will include approximately 500 patients with moderate to severe COPD from approximately 50 sites (including hospitals and GP practices) in Germany. Patients eligible for TRIXEO therapy may be enrolled by their treating physicians. The decision to treat with TRIXEO must be independent of the study and made by the treating physician according to the patients' medical need and local routine clinical practice. Patients' data will be collected for 12 months after starting therapy with TRIXEO.

Demographic and clinical data will be extracted from patients' health care records. Patient reported outcomes will be collected remotely by asking patients to answer questionnaires on health status and HRQoL, physical activity, sleep quality, treatment satisfaction, and inhaled medication adherence through electronic surveys.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed COPD
* Having been prescribed treatment with TRIXEO according to label and local market reimbursement criteria
* Patients must be able and willing to read and to comprehend written instructions, and to comprehend and complete the questionnaires required by the protocol
* After full explanation, patients must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* COPD due to α-1 antitrypsin deficiency
* Previous treatment with any other triple fixed-dose combination during screening
* Hospitalisation due to COPD exacerbation within the last 4 weeks prior to enrolment
* Pregnancy or lactation period
* Participation in an observational trial that might, in the investigator's opinion, influence the assessment for the current study, or participation in a randomised clinical trial in the last 30 days.
* Patient still recovering from Covid-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this study is patients with moderate to severe COPD and who have been prescribed TRIXEO therapy in the primary care or hospital care setting may be enrolled in this study. Patients meeting all the inclusion criteria and none of the exclusion criteria may be enrolled by their physician.
  The decision to start treatment with TRIXEO has to be made by the treating physician according to the subjects' medical need and a positive benefit/risk balance. The decision is not part of the study, lies with the treating physician and is taken according to the standard of current best medical practice and national guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in COPD Assessment Test (CAT) score after 3 months treatment | 3 months
  To describe the change in COPD health status after 3 months of treatment vs baseline in eligible COPD patients initiated with TRIXEO treatment

SECONDARY OUTCOMES:
Change from baseline in CAT score after 1, 6 and 12 months treatment | 12 months
  Describe change in COPD health status after 1, 6 and 12 months of treatment vs baseline in eligible COPD patients initiated with TRIXEO treatment
Change from baseline in St George's Respiratory Questionnaire (SGRQ) score after 3 and 12 months treatment | 12 months
  Describe change in health-related quality of life (HRQL) after 3 and 12 months vs baseline in eligible COPD patients initiated with TRIXEO treatment
Change from baseline in activity limitations, measured by CAT activity question/domain, after 1, 3 and 12 months of treatment | 12 months
  Describe change in physical activity and activity limitation at 1, 3, and 12 months of treatment vs baseline in eligible COPD patients initiated with TRIXEO treatment
Change from baseline in activity limitations, measured by SGRQ activity question/domain, after 3 and 12 months of treatment | 12 months
  Describe change in physical activity and activity limitation at 1, 3, and 12 months of treatment vs baseline in eligible COPD patients initiated with TRIXEO treatment
IQVIA Treatment Satisfaction Questionnaire for Medication (TSQM)© scores at baseline, 3 and 12 months | 12 months
  Describe change in patient satisfaction with their inhalation device after 3 and 12 months vs baseline in eligible COPD patients initiated with TRIXEO treatment
Change from baseline in exacerbation rate (moderate, severe) after 6 and 12 months of treatment | 12 months
  Describe change in physician-reported exacerbation rate (moderate and severe exacerbations) after 6 and 12 months vs baseline in eligible COPD patients initiated with TRIXEO treatment

CONTACTS AND LOCATIONS:
Locations (52):
- Germany (52):
  - Research Site, Böblingen, Germany
  - Research Site, Doerfles-Esbach, Germany
  - Research Site, Fürstenwalde, Germany
  - Research Site, Marburrg, Germany
  - Research Site, Auerbach
  - Research Site, Augsburg
  - Research Site, Bad Neustadt A.d. Saale
  - Research Site, Bayreuth
  - Research Site, Beelitz
  - Research Site, Berlin
  - Research Site, Biberach
  - Research Site, Bremen
  - Research Site, Cottbus
  - Research Site, Darmstadt
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Echterdingen
  - Research Site, Ehringshausen
  - Research Site, Filderstadt
  - Research Site, Flensburg
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Fürth
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hattingen
  - Research Site, Ibbenbueren
  - Research Site, Kronach
  - Research Site, Laage
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, Markkleeberg
  - Research Site, Nuremberg
  - Research Site, Peißenberg
  - Research Site, Potsdam
  - Research Site, Rathenow
  - Research Site, Rendsburg
  - Research Site, Rosenheim
  - Research Site, Rostock
  - Research Site, Roth
  - Research Site, Saalfeld
  - Research Site, Saarlouis
  - Research Site, Schleswig
  - Research Site, Teuchern
  - Research Site, Treuchtlingen
  - Research Site, Ulm
  - Research Site, Weißenburg
  - Research Site, Wiesbaden
  - Research Site, Wilhelmshaven
  - Research Site, Witten
  - Research Site, Würzburg
  - Research Site, Zirndorf

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D5980R00037_CSR Synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00037&attachmentIdentifier=43f18fe9-9e10-47c1-99ab-25d8e9b538da&fileName=D5980R00037_CSR_Synopsis_redacted.pdf&versionIdentifier=